CLINICAL TRIAL: NCT02021773
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Parallel Group, Multi-dose Study Comparing the Efficacy and Safety of Subcutaneous LBR-101 With Placebo for the Preventive Treatment of Chronic Migraine
Brief Title: Assessment of LBR-101 In Chronic Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LBR-101-021
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Results first posted 2021-11-01 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Chronic Migraine
Keywords: Headache; Migraine; Chronic Migraine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- LBR-101 High Dose (Experimental): Subcutaneous High Dose LBR-101 Administered Monthly x 3
  Interventions: Drug: LBR-101 High Dose
- LBR-101 Low Dose (Experimental): Subcutaneous Low Dose LBR-101 Administered Monthly x 3
  Interventions: Drug: LBR-101 Low Dose
- Placebo (Placebo Comparator): Subcutaneous Placebo Administered Monthly x 3
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LBR-101 High Dose — Subcutaneously Administered LBR-101 Monthly x 3
  Other Names: Fremanezumab
  Arms: LBR-101 High Dose
Drug: LBR-101 Low Dose — Subcutaneously Administered LBR-101 Monthly x 3
  Other Names: Fremanezumab
  Arms: LBR-101 Low Dose
Drug: Placebo — Subcutaneously Administered Placebo (Vehicle) Monthly x 3
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether monthly subcutaneous administration of LBR-101 (fremanezumab) is safe and provides migraine prevention in patients with chronic migraine.

DETAILED DESCRIPTION:
Two distinct doses of subcutaneous LBR-101 (fremanezumab) administered monthly will be compared to placebo for safety and efficacy. The mean change from baseline in the number of cumulative headache hours measured at the 28-day period ending with week 12.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 65 years of age.
* A signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study including any known and potential risks and available alternative treatments.
* Chronic migraine meeting the diagnostic criteria listed in the International Classification of Headache Disorders (ICHD-III beta version, 2013)
* Body Mass Index (BMI) of 17.5 to 37.5 kg/m2, and a total body weight between 50 kg and 120 kg inclusive.
* Demonstrated compliance with the electronic headache diary during the run-in period headache data on a minimum of 22/28 days (80% diary compliance)

Exclusion Criteria:

* Onset of chronic migraine after the age of 50 years.
* Subject has received onabotulinum toxin A for migraine or for any medical or cosmetic reasons requiring injections in the head, face, or neck during the 6 months prior to study entry.
* Subject is using medications containing opioids (including codeine) or barbiturates (including Fiorinal®, Fioricet®, or any other combination containing butalbital) on more than 4 days per month for the treatment of migraine or for any other reason.
* Failed > 2 medication categories or > 3 preventive medications (within two medication categories) due to lack of efficacy for prophylactic treatment of episodic or chronic migraine after an adequate therapeutic trial
* Treatment with an investigational drug or device within 30 days of study entry or any prior exposure to a monoclonal antibody targeting the CGRP pathway.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2015-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (57):
- United States (57):
  - Teva Investigational Site 145, Gilbert, Arizona
  - Teva Investigational Site 130, Phoenix, Arizona
  - Teva Investigational Site 117, Scottsdale, Arizona
  - Teva Investigational Site 161, Anaheim, California
  - Teva Investigational Site 116, Fullerton, California
  - Teva Investigational Site 119, Long Beach, California
  - Teva Investigational Site 146, Oceanside, California
  - Teva Investigational Site 113, San Francisco, California
  - Teva Investigational Site 108, Stanford, California
  - Teva Investigational Site 112, Walnut Creek, California
  - Teva Investigational Site 132, Boulder, Colorado
  - Teva Investigational Site 162, Stamford, Connecticut
  - Teva Investigational Site 143, DeLand, Florida
  - Teva Investigational Site 137, Hialeah, Florida
  - Teva Investigational Site 101, Jacksonville, Florida
  - Teva Investigational Site 166, Jacksonville, Florida
  - Teva Investigational Site 129, Maitland, Florida
  - Teva Investigational Site 167, Orlando, Florida
  - Teva Investigational Site 139, Ormond Beach, Florida
  - Teva Investigational Site 140, Port Orange, Florida
  - Teva Investigational Site 149, Atlanta, Georgia
  - Teva Investigational Site 164, Decatur, Georgia
  - Teva Investigational Site 134, Douglasville, Georgia
  - Teva Investigational Site 125, Evansville, Indiana
  - Teva Investigational Site 133, Lenexa, Kansas
  - Teva Investigational Site 135, Brockton, Massachusetts
  - Teva Investigational Site 124, New Bedford, Massachusetts
  - Teva Investigational Site 151, Springfield, Massachusetts
  - Teva Investigational Site 109, Watertown, Massachusetts
  - Teva Investigational Site 115, Worcester, Massachusetts
  - Teva Investigational Site 110, Ann Arbor, Michigan
  - Teva Investigational Site 114, Kalamazoo, Michigan
  - Teva Investigational Site 150, Golden Valley, Minnesota
  - Teva Investigational Site 152, Kansas City, Missouri
  - Teva Investigational Site 107, Springfield, Missouri
  - Teva Investigational Site 104, St Louis, Missouri
  - Teva Investigational Site 148, Reno, Nevada
  - Teva Investigational Site 105, The Bronx, New York
  - Teva Investigational Site 131, Greensboro, North Carolina
  - Teva Investigational Site 118, Raleigh, North Carolina
  - Teva Investigational Site 168, Winston-Salem, North Carolina
  - Teva Investigational Site 122, Canton, Ohio
  - Teva Investigational Site 141, Cincinnati, Ohio
  - Teva Investigational Site 142, Cincinnati, Ohio
  - Teva Investigational Site 155, Cleveland, Ohio
  - Teva Investigational Site 102, Columbus, Ohio
  - Teva Investigational Site 127, Oklahoma City, Oklahoma
  - Teva Investigational Site 111, Philadelphia, Pennsylvania
  - Teva Investigational Site 120, Goose Creek, South Carolina
  - Teva Investigational Site 153, Bristol, Tennessee
  - Teva Investigational Site 126, Memphis, Tennessee
  - Teva Investigational Site 154, Nashville, Tennessee
  - Teva Investigational Site 128, Arlington, Texas
  - Teva Investigational Site 121, Austin, Texas
  - Teva Investigational Site 136, Austin, Texas
  - Teva Investigational Site 123, Charlottesville, Virginia
  - Teva Investigational Site 144, Roanoke, Virginia

REFERENCES:
- [Derived] VanderPluym J, Dodick DW, Lipton RB, Ma Y, Loupe PS, Bigal ME. Fremanezumab for preventive treatment of migraine: Functional status on headache-free days. Neurology. 2018 Sep 18;91(12):e1152-e1165. doi: 10.1212/01.wnl.0000544321.19316.40. Epub 2018 Aug 17. PMID 30120138
- [Derived] Halker Singh RB, Aycardi E, Bigal ME, Loupe PS, McDonald M, Dodick DW. Sustained reductions in migraine days, moderate-to-severe headache days and days with acute medication use for HFEM and CM patients taking fremanezumab: Post-hoc analyses from phase 2 trials. Cephalalgia. 2019 Jan;39(1):52-60. doi: 10.1177/0333102418772585. Epub 2018 May 3. PMID 29722276
- [Derived] Cohen JM, Dodick DW, Yang R, Newman LC, Li T, Aycardi E, Bigal ME. Fremanezumab as Add-On Treatment for Patients Treated With Other Migraine Preventive Medicines. Headache. 2017 Oct;57(9):1375-1384. doi: 10.1111/head.13156. Epub 2017 Sep 1. PMID 28862758
- [Derived] Bigal ME, Edvinsson L, Rapoport AM, Lipton RB, Spierings EL, Diener HC, Burstein R, Loupe PS, Ma Y, Yang R, Silberstein SD. Safety, tolerability, and efficacy of TEV-48125 for preventive treatment of chronic migraine: a multicentre, randomised, double-blind, placebo-controlled, phase 2b study. Lancet Neurol. 2015 Nov;14(11):1091-100. doi: 10.1016/S1474-4422(15)00245-8. Epub 2015 Sep 30. PMID 26432181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 264 participants with chronic migraine were enrolled in the study.
Pre-assignment Details: Participants were assigned to receive either monthly subcutaneous administration of 900 mg of LBR-101 (fremanezumab), subcutaneous loading dose of 675 mg of LBR-101 (fremanezumab) followed by monthly subcutaneous doses of 225 mg of LBR-101 (fremanezumab), or monthly subcutaneous doses of placebo.
Groups:
- Placebo: Participants received subcutaneous placebo injections at one visit per month for three months (Day 1/week 0, Day 29/week 4, and Day 57/week 8).
- LBR-101 Low Dose: Participants received one subcutaneous loading dose of 675 mg LBR-101 (fremanezumab) on Day 1/week 0 followed by one subcutaneous dose of 225 mg LBR-101 (fremanezumab) once per month for two months (Day 29/week 4 and Day 57/week 8).
- LBR-101 High Dose: Participants received one subcutaneous dose of 900 mg LBR-101 (fremanezumab) once per month for three months (Day 1/week 0, Day 29/week 4, and Day 57/week 8).
Period: Overall Study
Arm/Group | Placebo | LBR-101 Low Dose | LBR-101 High Dose
Started (All randomized participants) | 89 | 88 | 87
Safety Analysis Set (Safety set: all participants who received at least one dose of study drug) | 89 | 88 | 86
Intent-to-treat (ITT) (All participants evaluable for efficacy) | 89 | 87 | 85
Completed | 77 | 72 | 76
Not Completed | 12 | 16 | 11
Not completed — Adverse Event | 1 | 4 | 3
Not completed — Lack of Efficacy | 2 | 2 | 2
Not completed — Protocol Violation | 2 | 3 | 1
Not completed — Withdrawal by Subject | 3 | 4 | 5
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Reason not specified | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LBR-101 Low Dose | LBR-101 High Dose | Total
Number analyzed (Participants) | 89 | 88 | 87 | 264
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (11.46) | 40.0 (11.56) | 41.5 (12.89) | 40.8 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 76 | 75 | 227
  Male | 13 | 12 | 12 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 14 | 10 | 35
  Not Hispanic or Latino | 78 | 74 | 77 | 229
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 12 | 9 | 30
  White | 76 | 70 | 73 | 219
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 5 | 14
Years of migraine [Mean (Standard Deviation); unit: Years] | 20.4 (13.14) | 15.8 (11.22) | 18.8 (12.2) | 18.3 (12.32)
Preventive Medication Use [Count of Participants; unit: Participants] — Participants reported preventive migraine medication use at the time of randomization
  Participants
    Yes | 38 | 35 | 33 | 106
    No | 51 | 53 | 54 | 158

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Number of Monthly Cumulative Headache Hours of Any Severity on Headache Days Relative to the 28-day Post-treatment Period Ending With Week 12
Description: A headache day was defined as when at least 1 of the following situations occurred: A calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache of any severity or the participant used acute migraine medication (triptans and ergot compounds) to treat a headache. This calculation was defined as the change from baseline in the number of hours with headache of any severity during the 28-day post treatment period ending at week 12. Headache severity was rated daily by the participant as either no pain, mild, moderate, or severe.
Time Frame: Baseline to week 12
Population: Intent-to-treat (ITT) population includes all randomized participants who received at least one dose of study drug and obtained at least one endpoint measurement.
Measure: Least Squares Mean (Standard Error); unit: Number of monthly headache hours
Arm/Group | Placebo | LBR-101 Low Dose | LBR-101 High Dose
Number analyzed (Participants) | 89 | 87 | 85
Number of monthly headache hours | -37.10 (8.42) | -59.84 (8.62) | -67.51 (8.61)
Statistical Analysis 1: Comparison: Placebo vs LBR-101 Low Dose; Test type: Superiority; p = 0.0386, Mixed Models Analysis — The threshold for statistical significance was p = .05; Mean Difference (Final Values) = -22.74, 95% CI 2-sided [-44.28 to -1.21], Standard Error of Mean 10.937
Statistical Analysis 2: Comparison: Placebo vs LBR-101 High Dose; Test type: Superiority; p = 0.0057, Mixed Models Analysis — The threshold for statistical significance was p = .05; Mean Difference (Final Values) = -30.41, 95% CI 2-sided [-51.88 to -8.95], Standard Error of Mean 10.90

2. Primary Outcome: Number of Participants With at Least One Adverse Event
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Relationship of AE to treatment was determined by the Investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent the previously listed serious outcomes. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline to week 12
Population: Safety analysis set included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | LBR-101 Low Dose | LBR-101 High Dose
Number analyzed (Participants) | 89 | 88 | 86
Participants | 36 | 47 | 41

3. Secondary Outcome: Mean Change From Baseline in the Number of Headache Days of at Least Moderate Severity Relative to the 28-day Post-treatment Period Ending With Week 12
Description: A headache day was defined as when at least 1 of the following situations occurred: A calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache of any severity or the participant used acute migraine medication (triptans and ergot compounds) to treat a headache. This calculation was defined as the change from baseline in the number of headache days of at least moderate severity during the 28-day post treatment period ending at week 12. Headache severity was rated daily by the participant as either no pain, mild, moderate, or severe.
Time Frame: Baseline to week 12
Population: Intent-to-treat (ITT) population includes all randomized participants who received at least one dose of study medication and obtained at least one endpoint measurement.
Measure: Least Squares Mean (Standard Error); unit: Number of headache days
Arm/Group | Placebo | LBR-101 Low Dose | LBR-101 High Dose
Number analyzed (Participants) | 89 | 87 | 85
Number of headache days | -4.20 (0.67) | -6.04 (0.687) | -6.16 (0.686)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks after first dose of treatment drug.
Description: Safety analysis set included all participants that received at least one dose of study treatment.
Arm/Group | Placebo | LBR-101 Low Dose | LBR-101 High Dose
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/88 | 0/86
Serious Adverse Events (participants affected / at risk) | 1/89 | 1/88 | 2/86
Other Adverse Events (participants affected / at risk) | 3/89 | 6/88 | 8/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=89) | LBR-101 Low Dose (N=88) | LBR-101 High Dose (N=86)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=89) | LBR-101 Low Dose (N=88) | LBR-101 High Dose (N=86)
Injection site pain (General disorders) | 3 (5) | 6 (8) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.